CLINICAL TRIAL: NCT07380763
Title: Comparison of Peri-intubation Oxygenation Values and Complications in Patients Intubated With the Delayed Sequential Intubation (DSI) Versus Rapid Sequence Intubation (RSI) Protocols
Brief Title: Comparison of Peri-intubation Oxygenation Values and Complications in Patients Intubated With the Delayed Versus Rapid Sequence Intubation Protocols
Acronym: DSI vs RSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Utku Murat Kalafat, Associate Professor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4975; 2024-KAEK-18 (Other: İSTANBUL HAYDARPAŞA NUMUNE EĞİTİM VE ARAŞTIRMA HASTANESİ KLİNİK ARAŞTIRMALAR ETİK KURULU)
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Delayed Sequence Intubation; Rapid Sequence Induction and Intubation; Intubation; Intubation Complications; Intubation, Endotracheal
Keywords: delayed sequence intubation; rapid sequence intubation; RSI; DSI
MeSH Terms: interventions — Rapid Sequence Induction and Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Sequence Intubation (Experimental)
  Interventions: Procedure: Delayed Sequence Intubation
- Rapid Sequence Intubation (Active Comparator)
  Interventions: Procedure: Rapid Sequence Intubation

INTERVENTIONS:
Procedure: Delayed Sequence Intubation — Patients assigned to the Delayed Sequence Intubation (DSI) protocol will receive an initial dose of 1 mg/kg ketamine. Titrated additional doses of 0.5 mg/kg will be administered until 'adequate sedation/dissociation' is achieved, ensuring the preservation of airway reflexes and spontaneous respiration. Subsequently, 'preoxygenation' will be performed for 3 minutes with 'appropriate positioning,' using a non-rebreather mask or bag-valve-mask combined with a nasal cannula delivering maximum oxygen flow (10-15 L/min). Following the induction of paralysis with an intravenous push of rocuronium (1 mg/kg), endotracheal intubation will be performed using direct laryngoscopy. Throughout the protocol, relevant physiological parameters will be recorded on the study data form by a designated physician.
  Arms: Delayed Sequence Intubation
Procedure: Rapid Sequence Intubation — Patients assigned to the Rapid Sequence Intubation (RSI) protocol will receive 'preoxygenation' for 3 minutes using a non-rebreather mask (NRM) or bag-valve-mask (BVM) combined with a nasal cannula delivering maximum oxygen flow (10-15 L/min), following the necessary preparation period. Subsequently, appropriate sedation and paralysis will be achieved through the sequential administration of intravenous (IV) ketamine (1 mg/kg push) and rocuronium (1 mg/kg IV push). Following induction, endotracheal intubation will be performed via direct laryngoscopy. Throughout the protocol, relevant physiological parameters will be recorded on the study data form by a designated physician
  Arms: Rapid Sequence Intubation

SUMMARY:
This study compares two different methods of helping patients breathe by placing a tube in their airway (intubation) in an emergency setting. These methods are called Rapid Sequence Intubation (RSI) and Delayed Sequence Intubation (DSI).

The study focuses on adult patients who are still breathing on their own but need a breathing tube for medical reasons not related to an injury (non-trauma).

The main goal of the research is to compare:

* Oxygen levels before and after the procedure.
* The patient's vital signs (such as heart rate and blood pressure).
* The number of attempts needed to successfully place the tube and the time the procedure takes.
* Blood gas results and any complications that occur during or shortly after the procedure.
* Early survival (mortality) rates.

While there are previous studies on trauma patients or small observational reports, there is currently no large-scale, multicenter randomized controlled trial that includes all non-trauma adult patients.

What makes this study unique? Confirmation of Tube Placement: Researchers will use a specific measurement called end-tidal CO2 (etCO2) to confirm the tube is in the right place, a method not used in similar previous studies.

Assessing Difficulty: This study will use the Cormack-Lehane classification system to measure how difficult the intubation was for each patient.

Standardization: For the first time, breathing machine (ventilator) settings will be standardized for all patients in this type of study.

Real-World Practice: By involving all emergency department physicians as practitioners, the study aims to show how these methods work across a wide range of medical teams.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Presence of spontaneous breathing.
3. No prediction of a difficult airway prior to intubation.
4. Requirement for advanced airway management.
5. Not in cardiac arrest.
6. Decided to intubate due to non-traumatic etiologies.
7. Planned intubation using ketamine for sedation and rocuronium for paralysis.
8. Decision to intubate due to one of the following clinical conditions:

   1. Acute Respiratory Failure: Patients with hypoxic or hypercapnic respiratory failure where adequate oxygenation cannot be achieved despite non-invasive ventilation.
   2. Inability to Protect the Airway: Altered level of consciousness or increased risk of pulmonary aspiration due to conditions such as upper gastrointestinal bleeding, ileus, volvulus, gastric outlet obstruction, hypersalivation, or hyperemesis.
   3. Shock States: Patients in any state of shock (hypovolemic, distributive, cardiogenic, obstructive) exhibiting severe altered mental status or declining respiratory status.
   4. Neuroprotection: Need to terminate ongoing seizures resistant to medical therapy (status epilepticus), or situations requiring strict control of arterial carbon dioxide (PaCO₂) levels to manage increased intracranial pressure (ICP) in non-traumatic conditions (such as intracranial hemorrhage or severe encephalopathy).
9. Obtaining informed consent from the patient or their legally authorized representative.

Exclusion Criteria:

1. Aged under 18 years.
2. Pregnancy.
3. Refusal to provide informed consent.
4. Cardiac arrest prior to intubation.
5. Anticipated difficult airway.
6. Intubation required due to traumatic etiologies.
7. Missing or incomplete patient data.
8. Patients assigned to the DSI protocol but for whom the decision to intubate was rescinded due to clinical improvement during the preoxygenation phase.
9. Use of a sedative agent other than ketamine for the RSI protocol.
10. Intubations performed by practitioners who have not received study-specific training on DSI and RSI protocols.
11. Duplicate enrollment due to recurrent presentations during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Procedure-Related Adverse Events | During and 1 hours after intubation
  Hypoxia(Spo2<90), hypotension (systolic blood pressure <90mmHg or blood pressure drop >20mmg after intiation of intubation protocol), orogastric intubation, cardiac arrest, orolaryngeal trauma, aspiration of orogastric fluid is accepted as procedure-related adverse events
Mean Peripheral Oxygen Saturation (SpO2) | Hospital admission, Intubation decision, Protocol start (0 min), Minutes 1, 2, 3 of protocol, During blade insertion, 1 minute post-intubation, and 5 minutes post-intubation
  Spo2 levels at admission, when intubation decision made, Spo2 level upon commencement of the intubation protocol(0-min); Spo2 level at 1st minute, 2nd minute, 3rd minute of intubation protocol, during blade passes incisor teeth, 1 minutes after intubation, 5 minutes after intubation wil be recorded
Mean Arterial Blood pH Levels | Hospital admission, At the time of intubation decision, and 15 minutes post-intubation.
  Evaluation of acid-base status.
Mean Partial Pressure of Carbon Dioxide (PaCO2) | Hospital admission, At the time of intubation decision, and 15 minutes post-intubation.
  Measure of carbon dioxide in arterial blood.
Mean Arterial Bicarbonate (HCO3) Concentration | Hospital admission, At the time of intubation decision, and 15 minutes post-intubation.
  Measure of bicarbonate in arterial blood.
Mean Base Excess (BE) Levels | Hospital admission, At the time of intubation decision, and 15 minutes post-intubation.
  Measure of base excess in arterial blood.
Mean Arterial Lactate Concentration | Hospital admission, At the time of intubation decision, and 15 minutes post-intubation.
  Measure of lactate in arterial blood.
First Hour Mortality | 1 hour later intubation
  Death from any cause within 60 minutes following the intubation attempt.
28th day mortality | 28 days after intubation
  All-cause mortality recorded during the first 28 days after enrollment.

SECONDARY OUTCOMES:
Number of intubation attempts | During the procedure (from the start of the intubation attempt until confirmation of tube placement).
  From the initiation of intubation until successful intubation is achieved.
Intubation Duration | During the procedure (from the start of the intubation attempt until confirmation of tube placement).
  Time from the laryngoscope blade passing the incisors until successful ETT placement.

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Basaksehir Cam and Sakura City Hospital, Istanbul, Istanbul
  - İstanbul Haseki Training and Research Hospital, Istanbul
  - Kanuni Sultan Süleyman Research and Training Hospital, Istanbul
  - Şişli Hamidiye Etfal Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
After publication and upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months and ending 36 months after article publication.
Access Criteria: Requests for data should be directed to the principal investigator. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Deyerle WM. Symposium on new surgical approaches. Clin Orthop Relat Res. 1973 Mar-Apr;(91):2. No abstract available. PMID 4703154
- [Background] Weingart SD, Trueger NS, Wong N, Scofi J, Singh N, Rudolph SS. Delayed sequence intubation: a prospective observational study. Ann Emerg Med. 2015 Apr;65(4):349-55. doi: 10.1016/j.annemergmed.2014.09.025. Epub 2014 Oct 23. PMID 25447559
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Stanke L, Nakajima S, Zimmerman LH, Collopy K, Fales C, Powers W 4th. Hemodynamic Effects of Ketamine Versus Etomidate for Prehospital Rapid Sequence Intubation. Air Med J. 2021 Sep-Oct;40(5):312-316. doi: 10.1016/j.amj.2021.05.009. Epub 2021 Jul 2. PMID 34535237
- [Background] Sehdev RS, Symmons DA, Kindl K. Ketamine for rapid sequence induction in patients with head injury in the emergency department. Emerg Med Australas. 2006 Feb;18(1):37-44. doi: 10.1111/j.1742-6723.2006.00802.x. PMID 16454773